CLINICAL TRIAL: NCT03584984
Title: Alveolar Ridge Preservation in Mandibular Molars Using Mixture of Autogenous Bone & Anorganic Bovine Bone (ABB) Versus Anorganic Bovine Bone Alone Versus Absorbent Gelatin Sponge
Brief Title: Autogenous Bone Mixed With Xenograft Versus Xenograft Alone Versus Absorbent Gelatin Sponge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mohammed Al-esawy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2807
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Bone Resorption; Alveolar Bone Loss; Alveolar Bone Resorption; Bone Graft Failure
MeSH Terms: conditions — Bone Resorption; Alveolar Bone Loss | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mixture of Autogenous bone & Anorganic Bovine Bone (ABB) (Experimental): socket preservation with a mixture of autogenous bone graft acquired at the time of extraction mixed with a 50:50 ratio of Anorganic bovine bone
  Interventions: Procedure: Mixture of Autogenous bone & Anorganic Bovine Bone (ABB)
- Anorganic bovine bone graft (ABB) (Active Comparator): filling the extraction socket with ABB graft
  Interventions: Procedure: Anorganic Bovine Bone (ABB)
- Absorbable gelatin Sponge (Active Comparator): Filling the socket with an absorbable gelatin sponge
  Interventions: Procedure: Absorbable gelatin sponge

INTERVENTIONS:
Procedure: Mixture of Autogenous bone & Anorganic Bovine Bone (ABB) — Filling the socket with Mixing of autogenous bone graft and anorganic bovine bone in a 50:50 ratio
  Arms: Mixture of Autogenous bone & Anorganic Bovine Bone (ABB)
Procedure: Anorganic Bovine Bone (ABB) — Filling the socket with Anorganic bovine bone graft material only
  Arms: Anorganic bovine bone graft (ABB)
Procedure: Absorbable gelatin sponge — Filling the socket with an absorbable gelatin sponge foam pack
  Arms: Absorbable gelatin Sponge

SUMMARY:
Alveolar bone atrophy post-extraction has been well documented in the past years. normal healing event results in a minimal loss of vertical height (around 1 mm), but a substantial loss of width in the buccal-lingual plane (4-6 mm). Alveolar socket preservation is thought to deal with this issue as to prevent the loss of alveolar bone dimensions post extraction in the case of delayed implant placement

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hopeless mandibular molars indicated for extraction and implant placement in two stages that indicate socket preservation.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony Walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to a history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.
* Patients that refuse to be called back for implant placement post extraction.
* Patients that have exceeded bone resorption surrounding the tooth prior to extraction and require guided bone regeneration.
* Pregnant Females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Histomorphometrical bone analysis | 6 month post primary surgery
  histological bone core analysis

SECONDARY OUTCOMES:
Alveolar Bone marginal loss | 6 month post primary surgery
  CBCT measurements of marginal bone dimensional difference